CLINICAL TRIAL: NCT05764837
Title: The Immediate Effect of Posterior Chain Facilitation by Foam Rolling on Reactive Force Performance
Brief Title: Effectiveness of Foam Rolling on Selected Muscle Groups on Jumping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Harasimova foam rolling
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
Keywords: SMR; plyometrics; jumps over hurdles; posterior myofascial chain
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Facilitation of the posterior chain was performed by foam rolling (BLACKROLL, standard hardness), where the left lower limb was rolled first, then the right lower limb and finally the spinal erectors. Rolling was performed with a sense of the highest intensity and at a high rolling speed, across the full length and width of the muscle with both cranial and caudal rolling directions. Facilitation was performed on each muscle group in the distoproximal direction, in the order of:
  m. triceps surae, hamstrings, and m. gluteus maximus, with the proband attending to each muscle group for 30 s. Finally, bilateral facilitation of mm. erectores spinae in the lumbar and thoracic segments was performed, also for 30 s. The frequency of rolling was determined using a metronome at 1.5 Hz.
  Interventions: Other: Foam Rolling
- Control group (No Intervention): The control group of probands rested in a resting sitting position for 4 minutes after pre-tests, corresponding to the intervention period.

INTERVENTIONS:
Other: Foam Rolling — Foam rolling was performed for 4 minutes with the goal of affecting the entire myofascial posterior chain.
  Arms: Intervention group

SUMMARY:
An experiment elucidating the immediate effect of foam rolling of the posterior chain on reactive force performance that will represent multiple jumps over low obstacles. The measurements will be performed using the Optojump device, which will provide data on the time of foot contact with the ground and the jump height. The angles of the torso inclination to the vertical will also be measured during jumping.

DETAILED DESCRIPTION:
Fifteen women were selected for this experiment in the form of a randomized crossover study. Measurements were taken by leg jumps over 5 obstacles 125 cm apart. The pre-test was performed twice with a two-minute rest between each trial. Immediately after finishing the second trial, a randomly selected half of the probands performed posterior chain facilitation using a foam roller, facilitating first the left leg, then the right leg and finally spinal erectors. Rolling was performed with a sense of maximal intensity and at a high rolling speed across the full length and width of the muscle with both cranial and caudal rolling directions. Facilitation was performed on each muscle group in the distoproximal direction. Immediately following the intervention, a post-test was performed a total of 3 times, 1 minute after the intervention, 3 minutes after the intervention and 5 minutes after the intervention. The control measurement was performed the same way as the intervention, but the control group of probands rested in a resting sitting position for 4 minutes instead of foam rolling. After one week, a second measurement followed, where the original control group underwent the intervention measurement and vice versa.

The Optojump instrument (Microgate, Bolzano, Italy) was used to obtain the resistance and flight phase data. A video recording (GoPro HERO 9) was taken of the skipping procedure, from which photographs were taken over each obstacle at the moment of the greatest trunk tilt (the junction of the trochanter major and the external auditory canal exit) from the vertical axis.

ELIGIBILITY:
Inclusion Criteria:

* women
* age range 18-30 years
* regular training at least 3 times a week
* training with a minimum duration of 1.5 hours
* valid medical sports examination
* experience with jumping over hurdles
* having a problem with maintaining the physiological position of the torso when running

Exclusion Criteria:

* injuries
* acute illnesses
* chronic disease
* musculoskeletal limitations
* during convalescence

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Angles of inclination of the fuselage to the vertical. | 45 minutes
  Measurements were made using video recording (GoPro HERO 9), with 1080p resolution and a recording rate of 240fps. Subsequent analysis of torso tilt was performed in Kinovea, with video frames taken over each obstacle at the moment of greatest torso tilt relative to the vertical axis. Using the marked point above the trochanter major ossis femoris and the external auditory canal outlet, a trunk axis was created and used to measure the angle relative to the vertical axis.

SECONDARY OUTCOMES:
Foot to ground contact time. | 1 hour
  The Optojump instrument (Microgate, Bolzano, Italy) was used to acquire the resist phase data by means of laser shadowing. This data was transcribed into OptoJumpNext, from where it was transferred to an excel program and processed there.
Jump height. | 45 min
  The Optojump (Microgate, Bolzano, Italy) was also used to obtain the jump height data by using the resistance phase time, which is plugged into the formula, to obtain the jump height.

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr, Ph.D., Principal Investigator — Charles University, Faculty of physical education and sport
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No